CLINICAL TRIAL: NCT01604889
Title: A Phase 1/2 Randomized, Blinded, Placebo Controlled Study of Ipilimumab in Combination With Epacadostat or Placebo in Subjects With Unresectable or Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Further development of this compound with ipilimumab in the treatment of melanoma is no longer being pursued.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 24360-201
Record Dates: First submitted 2012-05-09; First posted 2012-05-24 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Melanoma
Keywords: Melanoma, Skin Cancer, Oncology
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasms | interventions — epacadostat; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Epacadostat 300 mg (Experimental): 300 mg twice daily (BID) in combination with ipilimumab
  Interventions: Drug: Epacadostat; Drug: ipilimumab
- Placebo in combination with ipilimumab (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: ipilimumab
- Epacadostat 25 mg (Experimental): 25 mg BID in combination with ipilimumab
  Interventions: Drug: Epacadostat; Drug: ipilimumab
- Epacadostat 50 mg (Experimental): 50 mg BID in combination with ipilimumab
  Interventions: Drug: Epacadostat; Drug: ipilimumab
- Epacadostat 75 mg (Experimental): 75 mg once a day (QD) in combination with ipilimumab
  Interventions: Drug: Epacadostat; Drug: ipilimumab

INTERVENTIONS:
Drug: Epacadostat
  Other Names: INCB024360
  Arms: Epacadostat 25 mg; Epacadostat 300 mg; Epacadostat 50 mg; Epacadostat 75 mg
Drug: Placebo — Placebo
  Arms: Placebo in combination with ipilimumab
Drug: ipilimumab — ipilimumab 3 mg/kg IV
  Arms: Placebo in combination with ipilimumab
Drug: ipilimumab — Doses to be determined following the completion of Phase I of the study
  Arms: Epacadostat 25 mg; Epacadostat 300 mg; Epacadostat 50 mg; Epacadostat 75 mg

SUMMARY:
The study design includes an open-label, dose escalation phase followed by a blinded, randomized phase, which combines epacadostat (an oral IDO1 inhibitor) with an approved therapy and compares to approved therapy plus placebo in metastatic melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 years or older with unresectable or metastatic melanoma.
* A life expectancy of >12 weeks.
* Laboratory ranges and medical criteria met, as defined within the protocol.
* Subject may have received more than 1 prior regimen of systematic treatment for unresectable or metastatic melanoma.
* For Phase 2 period of the study only, Subjects must have archival tumor tissue available and collected with the prior 6 months or accessible disease for pre-treatment, study biopsy.

Exclusion Criteria:

* Pregnant or nursing women.
* Current investigational trial participation with another investigational product or subjects who have received any anticancer medications within 21 days prior to screening (6 weeks for mitomycin-C or nitrosoureas.)
* Subjects receiving monoamine oxidase inhibitors (MAOI)s; subjects who have ever had Serotonin Syndrome after receiving one or more serotonergic drugs.
* Subjects who have received prior immune checkpoint inhibitors (eg anti-CTLA-4, anti-PD-1, anti- PD-L1 and others) who have had Grade 3 or 4 hepatotoxicity, immune colitis requiring infliximab, endocrine toxicity not controlled by replacement, any other Grade 4 immune adverse events (AEs) or ocular toxicity
* Subjects with protocol-specified active autoimmune process except vitiligo or thyroiditis.
* Subjects with concurrent conditions that would jeopardize the safety of the safety of the subject or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
Phase 1: Number of patients with adverse events as a measure of Safety and Tolerability. | Baseline and minimally every 3 weeks until discontinuation or death (estimated timeframe to be 29 months from first patient enrolled to last patient discontinued or dead).
Phase 2: Overall survival. | Measured every 4 weeks until the 50th death occurs, then follow-up is measured every 3 months (estimated timeframe to be 29 months from first patient enrolled to last patient death).

SECONDARY OUTCOMES:
Preliminary efficacy as assessed by tumor response. | Baseline and every nine weeks (3 cycles) thereafter (estimated timeframe is that each patient will be on study for 11 months).
Evaluation of progression free survival. | Measured every 4 weeks until the 50th death occurs, then follow-up is measured every 3 months (estimated timeframe is that patients will progress after 11 months).

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, M.D., Study Director — Incyte Corporation
Locations (7):
- United States (7):
  - Los Angeles, California
  - Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Gibney GT, Hamid O, Lutzky J, Olszanski AJ, Mitchell TC, Gajewski TF, Chmielowski B, Hanks BA, Zhao Y, Newton RC, Maleski J, Leopold L, Weber JS. Phase 1/2 study of epacadostat in combination with ipilimumab in patients with unresectable or metastatic melanoma. J Immunother Cancer. 2019 Mar 20;7(1):80. doi: 10.1186/s40425-019-0562-8. PMID 30894212